CLINICAL TRIAL: NCT05066399
Title: Fetal Cardiac Magnetic Resonance Imaging Using DUS Gating on 3T: Preliminary Experiences in Detection of CHD
Brief Title: Fetal Cardiac Magnetic Resonance in Detection of CHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Julian Alexander Luetkens, Principial Investigator, Senior Physician, University Hospital, Bonn
Other Study IDs: 523/20
Record Dates: First submitted 2021-09-22; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Congenital Heart Disease; Fetal Cardiac Disorder; Heart Defect, Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this clinical prospective study is to investigate the value of fetal cardiac magnetic resonance imaging using a new Doppler ultrasound based gating method for the detection of congenital heart desease.

ELIGIBILITY:
Inclusion Criteria:

* fetuses in third trimenon
* congenital heart defect suspected by obstetric ultrasound

Exclusion Criteria:

* pregnant women with contraindication for native MRI

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic (Department of Obstetrics and Prenatal Medicine, University Hospital Bonn, Germany), Prof. Dr. med. Annegret Geipel
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The number of heart defect characteristics detectable by DUS gated Cine MRI imaging | Up to 3 months after birth, cardiac MRI findings will be compared against fetal ultrasound gainst fetal ultrasounand against findings after birth (reference standard).
  DUS gated Cine imaging will be applied to detect characteristics of clinically suspected congenital heart defects.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Clinic for Diagnostic and Interventional Radiology, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No